CLINICAL TRIAL: NCT05201196
Title: Effects of Task Orientated Training on Dexterous Movement of Hand in Post Stroke Patients
Brief Title: Task Oriented Training in Post Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0235 Tahreem Zaman
Record Dates: First submitted 2021-11-08; First posted 2022-01-21 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: Stroke; Task; Training; Movement
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy (Active Comparator): Conventional physical therapy Muscle strengthening and Muscle Stretching, TENS.
  Interventions: Other: Conventional physical therapy
- Task Oriented Training (Experimental): Experimental group was given Task Oriented protocol including different task specific functional activities
  Interventions: Other: Task Oriented Training

INTERVENTIONS:
Other: Conventional physical therapy — Targeted muscle stretching and Strengthening (flexors, Extensors, abductors, internal and external rotators, of Shoulder, Elbow, forearm (supination & pronation) and hand 10 repetitions×1 set, 4 days/ week. Transcutaneous Electrical nerve Stimulation for 10-20 min, 4 days/ week. Total of 16 sessions were given each consisting of 45 mins.
  Arms: Conventional physical therapy
Other: Task Oriented Training — Experimental group was given Task oriented protocol including activities such as Table-top polishing, Arm cradling, Reach forward and pick-up or touch an object, Reached sideway to pick-up an object and transferring it to a table in front, Pouring
  ½ cup of water from a measuring pot into wide mouth glass held in opposite hand, Picking up pen from thumb and first two fingers, lifting a basket and placing it on the table 10 repetitions×1 set for each activity, 4-5days/week. Total of 16 sessions were given each consisting of 45 mins
  Arms: Task Oriented Training

SUMMARY:
This study will be observe the effect of Task-oriented training on the dexterous movements of hands in hemiparetic post-stroke patients. Patient will be recruited that meet the inclusion criteria, with unilateral hemiplegia referred by Neurophysician having stroke for the first time, between age 47-70 year, both males and females, score of spasticity for upper extremity (shoulder, elbow) below and equal 2 based on the Modified Ashworth Scale (MAS), ability to comprehend simple instructions (Mini-Mental State Examination with a minimum score > 24), Brunnstrom stages ≥ 4, not submitted to other upper-limb rehabilitation programs during the participation in this study. The individuals with recurrent stroke episodes and transient ischemic attack, other neurological diseases (Parkinson's disease, multiple sclerosis,), hemineglect, no sitting balance and comorbidities are excluded. Outcome measures used are FuglMeyer assessment scale (wrist and hand) and Wolf motor function test for upper extremity while Barthel index to assess the activities of daily living. All procedures will perform by taking informed consent. All Ethical standards for both patient and institution will be followed. After collecting data, will apply Shapiro Wilk test to check the normal distribution of data. For analysis use SPSS version 25

ELIGIBILITY:
Inclusion Criteria:

Unilateral hemiplegic stroke patients referred by Neuro-physician (both ischemic and hemiplegic stroke patients).

* Patient with first time stroke (within 6month of onset).
* Age between 45-70 years of age.
* Gender both male & females.
* Ability to comprehend simple instructions (Mini-Mental State Examination with a score of >24 ).
* Score of spasticity for upper extremity (shoulder, elbow) below and equal 2 based on the Modified Ashworth Scale (MAS).
* Motor recovery of upper limb Brunnstrom stages ≥ 4.
* Not participated to other upper-limb rehabilitation programs during the participation in this study.

Exclusion Criteria:

Recurrent stroke attacks, Transient ischemic attacks(TIA).

* Previous injury, disease, or contracture of the upper extremity and no sitting balance.
* Any comorbid neurological disease or condition such as multiple sclerosis, Parkinson disease, spinal cord injury, traumatic brain lesions, brain tumor, epilepsy, or dementia,
* Had Hemineglect phenomena.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Assessment (FMA-UE) | Pre treatment as baseline
  Fugl-Meyer upper extremity evaluates voluntary movement, reflex activity, grasp, and coordination. Performance is measured on with a 3-point ordinal scale (0 to 2), with a maximum score of 30 with sub score 10 for the wrist, 14 for the hand, and for coordination and speed of movement the score is 6
Fugl-Meyer Upper Extremity Assessment (FMA-UE) | Mid treatment after 3 weeks
  Fugl-Meyer upper extremity evaluates voluntary movement, reflex activity, grasp, and coordination. Performance is measured on with a 3-point ordinal scale (0 to 2), with a maximum score of 30 with sub score 10 for the wrist, 14 for the hand, and for coordination and speed of movement the score is 6
Fugl-Meyer Upper Extremity Assessment (FMA-UE) | Post treatment after 6 weeks
  Fugl-Meyer upper extremity evaluates voluntary movement, reflex activity, grasp, and coordination. Performance is measured on with a 3-point ordinal scale (0 to 2), with a maximum score of 30 with sub score 10 for the wrist, 14 for the hand, and for coordination and speed of movement the score is 6
Wolf Motor Function Test (WMFT) | Pre treatment as baseline
  Wolf motor function is a quantitative measure used for upper extremity motor ability using timed and functional tasks. It comprises of 15 function-based tasks and 2-strength based tasks. Maximum score is 75 and Lower scores are suggests low level of functioning. Time required for the task vary with individuals and usually 15-20 minutes
Wolf Motor Function Test (WMFT) | Mid treatment after 3 weeks
  Wolf motor function is a quantitative measure used for upper extremity motor ability using timed and functional tasks. It comprises of 15 function-based tasks and 2-strength based tasks. Maximum score is 75 and Lower scores are suggests low level of functioning. Time required for the task vary with individuals and usually 15-20 minutes
Wolf Motor Function Test (WMFT) | Post treatment after 6 weeks
  Wolf motor function is a quantitative measure used for upper extremity motor ability using timed and functional tasks. It comprises of 15 function-based tasks and 2-strength based tasks. Maximum score is 75 and Lower scores are suggests low level of functioning. Time required for the task vary with individuals and usually 15-20 minutes
Barthel Index | Pre treatment as baseline
  Barthel index include the data obtained from the patient's self-report, or from one of his attendants. It include 10-activities of daily living. These outcome measures are administrated at initial before 3 days of treatment, middle at 6 session and posttreatment
Barthel Index | Mid treatment after 3 weeks
  Barthel index include the data obtained from the patient's self-report, or from one of his attendants. It include 10-activities of daily living. These outcome measures are administrated at initial before 3 days of treatment, middle at 6 session and posttreatment
Barthel Index | Post treatment after 6 weeks
  Barthel index include the data obtained from the patient's self-report, or from one of his attendants. It include 10-activities of daily living. These outcome measures are administrated at initial before 3 days of treatment, middle at 6 session and posttreatment

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Pakistan(Punjab_, Pakistan

IPD SHARING:
Plan to Share IPD: No